CLINICAL TRIAL: NCT03608358
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 3 Trial to Evaluate the Safety and Efficacy of Dapagliflozin in Asian Subjects With T2DM and Inadequate Glycemic Control on Metformin and Saxagliptin (DS Navigation)
Brief Title: Safety and Efficacy of Dapagliflozin in Asian T2DM Subjects With Inadequate Glycemic Control on Metformin/Saxagliptin
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decided to stop commercialization of QTERNMet/Qtrilmet and to stop all related ongoing activities/studies for business reasons.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D1683C00008
Record Dates: First submitted 2018-07-11; First posted 2018-07-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: DPP-4 inhibitor; HbA1c; Incretin; Dapagliflozin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; saxagliptin; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dapagliflozin 10 mg (Experimental): Dapagliflozin 10 mg and dapagliflozin 5 mg placebo to match added to saxagliptin 5 mg and metformin
  Interventions: Drug: Dapagliflozin 10 mg; Drug: Dapagliflozin 5 mg placebo to match; Drug: Saxagliptin 5 mg; Drug: Metformin
- Dapagliflozin 5 mg (Experimental): Dapagliflozin 5 mg and dapagliflozin 10 mg placebo to match added to saxagliptin 5 mg and metformin
  Interventions: Drug: Dapagliflozin 5 mg; Drug: Dapagliflozin 10 mg placebo to match; Drug: Saxagliptin 5 mg; Drug: Metformin
- Placebo (Placebo Comparator): Dapagliflozin 5 mg placebo to match and dapagliflozin 10 mg placebo to match added to saxagliptin 5 mg and metformin
  Interventions: Drug: Dapagliflozin 10 mg placebo to match; Drug: Dapagliflozin 5 mg placebo to match; Drug: Saxagliptin 5 mg; Drug: Metformin

INTERVENTIONS:
Drug: Dapagliflozin 10 mg — 10 mg, oral tablet, once daily for 24 weeks of double-blind treatment period
  Arms: Dapagliflozin 10 mg
Drug: Dapagliflozin 5 mg — 5 mg, oral tablet, once daily for 24 weeks of double-blind treatment period
  Arms: Dapagliflozin 5 mg
Drug: Dapagliflozin 10 mg placebo to match — 10 mg, oral tablet, once daily for 24 weeks of double-blind treatment period
  Arms: Dapagliflozin 5 mg; Placebo
Drug: Dapagliflozin 5 mg placebo to match — 5 mg, oral tablet, once daily for 24 weeks of double-blind treatment period
  Arms: Dapagliflozin 10 mg; Placebo
Drug: Saxagliptin 5 mg — 5 mg, oral tablet, once daily for 24 weeks of double-blinded treatment period, and for 16 weeks of open-label treatment period in Stratum A or 8 weeks of open-label treatment period in Stratum B
Drug: Metformin — Stable dose of metformin immediate release/extended release (≥ 1500 mg/day or at a maximal tolerated dose) throughout the whole study period

SUMMARY:
This is a 24-week, multicenter, randomized, double-blind, double-dummy, placebo-controlled, parallel group, phase 3 study designed to evaluate if the safety and efficacy of dapagliflozin 5 mg or 10 mg added to saxagliptin 5 mg plus metformin is superior to placebo added to saxagliptin 5 mg plus metformin in reducing hemoglobin A1c (HbA1c).

DETAILED DESCRIPTION:
This study will be conducted in approximately 36 sites in Asian countries. Approximately 1004 subjects will be screened and 342 randomized. Prior to the screening, subjects of Stratum A should have a stable dose of metformin (≥1500 mg/day or a maximal tolerated dose) for at least 8 weeks. And subjects of Stratum B should have a stable dose of metformin (≥1500 mg/day or a maximal tolerated dose) AND a dipeptidyl peptidase-4 inhibitor at maximum approved dose for at least 8 weeks prior to the screening. Eligible subjects who complete the screening visit will enter the lead-in period, which includes open-label saxagliptin 5 mg and metformin treatment for 16 weeks in Stratum A or 8 weeks in Stratum B. At randomization visit, eligible subjects will be randomized into 1 of 3 treatment groups in a 1:1:1 ratio, receiving blinded dapagliflozin 5 mg, 10 mg or placebo plus metformin and saxagliptin 5 mg treatment for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent before participating in the study
2. Diagnosed with type 2 diabetes mellitus
3. Inadequate glycemic control defined as below:

   * HbA1c ≥ 8.0% and ≤ 11.5% for Stratum A and HbA1c ≥ 7.5% and ≤ 10.5% for Stratum B at screening visit
   * HbA1c ≥ 7.0 and ≤ 10.5% for both strata at Week -2 visit
4. Body mass index ≤ 40.0 kg/m^2

Exclusion Criteria:

1. Women of childbearing potential unable or unwilling to use acceptable birth control, or women who are pregnant or breastfeeding
2. History of diabetes insipidus and type 1 diabetes
3. History of diabetic ketoacidosis requiring medical intervention within 1 month prior to screening
4. Subjects with moderate to severe renal impairment (defined as estimate glomerular filtration rate calculated by the MDRD Formula < 60mL/min/1.73 m^2 or serum creatinine ≥ 1.5 mg/dL in males or ≥ 1.4 mg/dL in females) or end-stage renal disease
5. History of unstable or rapidly progressing renal disease
6. Subjects with significant hepatic disease or severe hepatic impairment, or positive serologic evidence of current infectious liver disease
7. Prohibited Treatment and Therapies

   * Administration of any anti-hyperglycemic therapy [other than metformin, or Dipeptidyl peptidase-4 (DPP-4) inhibitors] for more than 14 days (consecutive or not) during the 8 weeks prior to screening
   * Any use of Sodium glucose cotransporter 2 (SGLT2) inhibitor within 8 weeks prior to screening
   * Prescription and over-the-counter weight loss medications within 3 months prior to screening
   * Current treatment with potent cytochrome P450 3A4/5 inhibitors
8. Malignancy within 5 years of the screening
9. History of hemoglobinopathy
10. Hematuria (by microscopy) positive at screening visit
11. FPG > 270 mg/dL obtained at open-label period
12. An abnormal TSH value at screening will be further evaluated for free T4. Subjects with abnormal free T4 values will be excluded

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2020-08-04 (Actual); Study Completion 2020-08-04 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in HbA1c at Week 24 | Baseline to Week 24
  To compare the mean change from baseline in HbA1c achieved with dapagliflozin 5 mg or dapagliflozin 10 mg added to saxagliptin 5 mg plus metformin versus placebo added to saxagliptin 5 mg plus metformin after 24 weeks of oral administration of double-blind treatment

SECONDARY OUTCOMES:
Mean change from baseline in fasting plasma glucose (FPG) at Week 24 | Baseline to Week 24
  To compare the mean change from baseline in FPG achieved with dapagliflozin 5 mg or dapagliflozin 10 mg added to saxagliptin 5 mg plus metformin versus placebo added to saxagliptin 5 mg plus metformin after 24 weeks of oral administration of double-blind treatment
Mean change in 2-hour postprandial glucose during a meal tolerance test (2-hour MTT) at Week 24 | Baseline to Week 24
  To compare the mean change from baseline in 2-hour postprandial glucose from a meal tolerance test (2-hour MTT) achieved with dapagliflozin 5 mg or dapagliflozin 10 mg added to saxagliptin 5 mg plus metformin versus placebo added to saxagliptin 5 mg plus metformin after 24 weeks of oral administration of double-blind treatment
Mean change from baseline in total body weight at Week 24 | Baseline to Week 24
  To compare the mean change from baseline in total body weight achieved with dapagliflozin 5 mg or dapagliflozin 10 mg added to saxagliptin 5 mg plus metformin versus placebo added to saxagliptin 5 mg plus metformin after 24 weeks of oral administration of double-blind treatment
Percent of subjects achieving a therapeutic glycaemic response of HbA1c <7.0% at Week 24 | At week 24
  To compare the proportion of subjects achieving a therapeutic glycaemic response of HbA1c < 7.0% with dapagliflozin 5 mg or dapagliflozin 10 mg added to saxagliptin 5 mg plus metformin vs. placebo added to saxagliptin 5 mg plus metformin after 24 weeks of oral administration of double-blind treatment

CONTACTS AND LOCATIONS:
Overall Officials: Linong Ji, Professor, Principal Investigator — People's Hospital of Peking Universty
Locations (2):
- Research Site, Bangkok, Thailand
- Research Site, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Clinical Study Results on trialsummaries.com — https://www.trialsummaries.com/Study/StudyDetails?id=3235&tenant=MT_MED_9011

DOCUMENTS (2):
  • Study Protocol (2019-02-14): https://cdn.clinicaltrials.gov/large-docs/58/NCT03608358/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-29): https://cdn.clinicaltrials.gov/large-docs/58/NCT03608358/SAP_001.pdf